CLINICAL TRIAL: NCT06466499
Title: Non-pharmacological Treatment of Patients at Risk of Developing Persistent Posttraumatic Headache
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SashaRGN
Record Dates: First submitted 2024-06-06; First posted 2024-06-20 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Posttraumatic Headache
MeSH Terms: conditions — Post-Traumatic Headache

STUDY DESIGN:
Intervention Model Description: In the RCT measurements will be conducted three times; baseline, post intervention, and at six months follow-up.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): The control group will receive the standard treatment, which is oral and written information about the characteristic symptoms after head trauma, specific signals to be aware of, when to contact the general practitioner and guidance of gradual return to daily activities
- Intervention (Experimental): The intervention will cover an interdisciplinary 5-week program with sessions from both psychologists and physiotherapists. The psychologist sessions will focus on topics regarding cognitive behavioural therapy, psychoeducation, occupational rehabilitation and work activity. The physiotherapeutic sessions will include a combination of exercises on neck tensions, relaxation therapies and advises on, how to return gradually to daily activities (social, cognitive, and physical activities, such as reading, working by the computer, house cleaning, exercising, and going out with friends). Furthermore, patients will get exercise handouts to do at home between sessions.
  Both psychologist and physiotherapist sessions will be group-based with 6-8 patients in each group. Once every week, the groups receive psychologist sessions lasting 90 minutes and afterwards physiotherapist sessions of 60 minutes.
  Interventions: Behavioral: The intervention group

INTERVENTIONS:
Behavioral: The intervention group — Is described in arm
  Arms: Intervention

SUMMARY:
The goal of this mixed method study is to test and evaluate the effect of an early interdisciplinary non-pharmacological treatment of patients at risk of developing persistent posttraumatic headache in order to prevent the development of persistent posttraumatic headache and thereby, reduce persistency and improve the quality of life. Furthermore, to gain knowledge on and a deeper understanding of the patients' perspective and experience of the treatment.

The project consists of 3 sub studies:

1. A feasibility study; with the purpose of exploring the feasibility of an early non-pharmacological intervention for patients with persistent posttraumatic headache after mild traumatic brain injury.
2. An experimental design; a randomized controlled trial to evaluate the effect of the early non-pharmacological treatment.
3. A qualitative focus group interview study; to get a more nuanced knowledge of patients' experience with the non-pharmacological treatment related to post traumatic headache.

DETAILED DESCRIPTION:
The feasibility study will be performed prior to a randomized controlled trial and aim to assess the following: recruitment capability, data collection procedures and outcome measures, acceptability of the intervention, resources and ability to manage the study and intervention, and participant responses to the intervention.

Study population and recruitment The project will be conducted at the University Hospital of Southern Denmark. Patients will be recruited from the Emergency department. All patients hospitalized with mild traumatic brain injury (mTBI) will be asked to sign a statement of consent so the researcher is allowed to contact the patients for eligibility after three months. Participation in the study is voluntary. Patients will be informed about the feasibility nature of the study and included after oral consent. A neurological exam will be performed to assess final eligibility.

Patients are included 3-5 months after trauma and the intervention is initiated no later than six months after mTBI. In this study a sample size of 8 participants are chosen to assess feasibility.

Intervention The intervention will take place at the specialized Headache Clinic at the University Hospital of Southern Denmark. It will cover an interdisciplinary 5-week program with sessions from both psychologists and physiotherapists, all working at the Headache Clinic. The psychologist sessions will focus on topics regarding cognitive behavioural therapy, psychoeducation, occupational rehabilitation and work activity. The physiotherapeutic sessions will include a combination of exercises on neck tensions, relaxation therapies and advises on, how to return gradually to daily activities (social, cognitive, and physical activities, such as reading, working by the computer, house cleaning, exercising, and going out with friends). Furthermore, patients will get exercise handouts to do at home between sessions. Both psychologist and physiotherapist sessions will be group-based with 6-8 patients in each group. Once every week, the groups receive psychologist sessions lasting 90 minutes and afterwards physiotherapist sessions of 60 minutes.

The aim of the randomized controlled trial (RCT) is to investigate the effect of an early non-pharmacological treatment in patients at risk of developing persistent PTH. The null-hypothesis is that there is no difference between the groups, however the alternative hypothesis is that the intervention will result in reduced number of individuals with persistent headache 6 months after the trauma.

The overall preliminary set-up of the RCT study will be as in the feasibility study. Therefore recruitment, study population, measurements, intervention and standard treatment are as described above. The RCT measurements will be conducted three times; baseline, post intervention, and at six months follow-up.

The primary outcome is number of days with headache within the last week. There is no available reference of clinical trials regarding the group by time effect of non-pharmacological treatment on patients with persistent posttraumatic headache (PTH). In order to establish the premise for the sample size calculation, we therefore used results from studies on similar headache groups together with empirical clinical assumption. A study has shown that patients with persistent PTH of a moderate or severe intensity have an average of approximately 20 days per month, and we assume that approximately 20% reduction is clinically relevant. To detect at minimal clinically important difference (MICD) of 3,5 days, standard deviation (SD) (8.0) per month between the groups on two-sided significance level of 0.05 and power of 80%, it is required to enrol 83 patients in the intention to treat (ITT) population. We will include 52 participants in each group to account for dropouts.

Randomization will be performed after baseline measurements are collected using the web-based service Sealed envelope. Patients will be randomized (1:1) to receive either 5 weeks of interventional program or standard treatment. Block randomization (block sizes of 2, 4 and 6) are used and the principal researcher will be blinded to allocation.

Statistics Between group effects of the interventional program is assessed by mixed-effects models for repeated measurement, with a time factor for baseline, five weeks and six months. The model's residuals are tested for normal distribution and before conducting analyses, the variance homogeneity and assumption of linearity is investigated. To accommodate minor deviations from normally distributed data, robust estimation function will be applied. Analyses on the effects of the intervention is conducted according to the ITT principle, including all randomized patients irrespectively of withdrawal or drop-out. Subsequently, per protocol (PP) analyses is performed, including those patients from the intervention group who is compliant (attended ≥50% of the interventional sessions) compared with the patients from the control group. Missing data will be handled by multiple imputations, assuming that data is missing at random. Ten imputations are chosen as suitable. For hypothesis testing two-tailed tests is used and the significance level is <0.05 for all tests.

The qualitative focus group interview study will be conducted to gain knowledge of what it means to patients with PTH to participate in an early non-pharmacological intervention, with respect to perceived quality of life and self-management in daily activities after a head trauma.

Study participants and setting The participating patients are the same patients who attend the interventional program in the RCT study. Participants are at baseline asked if they will participate in an interview after the intervention. Participants, who agrees to the interview and signs an informed consent, will be invited for focus group interviews with health care professionals when intervention is complete. The researcher will through data saturation claim when enough participants have been interviewed to achieve research purpose. Data saturation refers to the point in the research process when no new information is discovered during the interviews. This redundancy signals to the researcher that interviews and thereby data collection may cease. There will be four focus group interviews conducted. Each focus group consists of five to six patients. All interviews will be performed at the University Hospital of Southern Denmark, after the 5-weeks intervention and the duration of the interviews are approximately 90 minutes.

Data collection The principal researcher and a researcher assistant will be facilitating the interviews, as this set-up provides capability for one to interact in the group conversations, while the other one notes interesting non-verbal interaction in the groups. A semi-structured interview guide will be developed prior to conducting the focus group interviews. Overall themes for the interview guide are; Thoughts about the intervention and how it affects their everyday life (illness mastery), changes in the general well-being after the intervention, changes in coping strategies, self-management, thoughts and feelings about the future.

Data analysis and interpretation The interviews will be audio recorded, verbatim transcribed and anonymized with pseudonyms by the principal investigator. Interview data are systematically entered into a qualitative data analyses software program for coding. The theoretical approach will be phenomenological-hermeneutic inspired by Paul Ricoeur's theory of narratives and interpretation. A three-phased interpretation process will be used; naïve reading which provides an initial overall impression of the data, structural analysis where the data are structured by units of meaning and units of significance providing themes and critical interpretation and discussion where the findings are interpreted and discussed with theory and research knowledge. This approach will allow the movement from individual perspective to a more general interpretation.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosed with acute posttraumatic headache
* Headache present for more than 15 days/month
* Must understand written and spoken Danish

Exclusion criteria:

* History of pre-existing primary or secondary headache
* Dementia or comorbidity with neurological disorders
* Psychiatric disorders
* Participants who cannot collaborate in relation to the intervention

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
Number of days with headache within the last week | 8 months
  The primary outcome is number of days with headache within the last week. Headache will be reported by a self-administered validated headache diary. Patients note every day if they experience any headache. The diary assesses days with headache graduated in intensity using a 1-3 scale (1= mild intensity and 3= severe intensity).

SECONDARY OUTCOMES:
Headache intensity | 8 months
  Secondary outcomes measures are headache intensity during the last 24 hours and intensity during the last week evaluated using a numeric rating scale. Two questions will be posed: "On a scale from 0 (equals no pain) to 10 (worst imaginable pain), please specify the degree of pain due to headache during the last 24 hours and "On a scale from 0 (equals no pain) to 10 (worst imaginable pain), please specify the degree of pain due to headache during the last week?"
Headache disability | 8 months
  To measure the severity of headache the Headache Impact Test (HIT6) is used. The questionnaire is a reliable and validated tool used to measure how big an impact headache has on patients' ability to function at work, at school, at home and in social relations.
Coping strategies | 8 months
  Coping strategies, will be measured by the Coping strategy Questionnaire (CSQ). The validated questionnaire includes six coping strategy subscales: Ignoring pain, reinterpretation of pain, diverting attention, coping self-statements, catastrophizing, praying/hoping, and two subscales for behavioral strategies: Increasing activity levels and increasing pain behaviors.
Mental health | 8 months
  Mental health will be measured by The 36-item Short Form Survey (SF-36).This is a reliable and validated instrument frequently used across different patient groups. The instrument consists of 36 items on perceived health-related quality of life, with answers divided into eight scales measuring health concepts: physical functioning, role physical, role emotional, social functioning, bodily pain, mental health, vitality and general health. All eight scales contribute in different proportions to the scoring of both physical and mental measures.
Physical functioning | 8 months
  Physical functioning will be measured by the SF-36
Emotional functioning | 8 months
  Emotional functioning will be measured by the SF-36
Number of sick leave days | 8 months
  This will be a customized question in the survey

IPD SHARING:
Plan to Share IPD: No